CLINICAL TRIAL: NCT04900597
Title: Effect of Blenderized Enteral Tube Feeds on Pediatric Upper Gastrointestinal Tract Physiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Bridget Hron, Staff Physician, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB-P00037093
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Enteral Feeding Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Elecare - Nourish - Real Foods Blends (Experimental): Elecare for first bolus, Nourish for second bolus, Real Foods Blends for third bolus
  Interventions: Other: Elecare Jr; Other: Nourish; Other: Real Foods Blends
- Nourish - Real Foods Blends - Elecare (Experimental): Nourish for first bolus, Real Foods Blends for second bolus, Elecare for first bolus
  Interventions: Other: Elecare Jr; Other: Nourish; Other: Real Foods Blends
- Real Foods Blends - Elecare - Nourish (Experimental): Real Foods Blends for first bolus, Elecare for second bolus, Nourish for third bolus
  Interventions: Other: Elecare Jr; Other: Nourish; Other: Real Foods Blends

INTERVENTIONS:
Other: Elecare Jr — Elecare Jr is a standard pediatric elemental formula
Other: Nourish — Nourish is a commercially prepared blenderized tube feed that is formulated for pediatric use
Other: Real Foods Blends — Real Foods Blends is a commercially prepared blenderized tube feed that is formulated for pediatric use

SUMMARY:
Blenderized diets consist of a wide range of table foods such as fruits, vegetables, meat and legumes, pureed in a blender and administered via gastrostomy tube. In a recent study, the investigators reported that children receiving blenderized feeds via gastrostomy had fewer total admissions and respiratory admissions, total emergency room visits, and improved gastrointestinal symptom scores compared to those fed formula. The goal of this project is to understand how these diets affect gastroesophageal reflux burden.

DETAILED DESCRIPTION:
The investigators hypothesize that rates of gastroesophageal reflux will be lower in blenderized diets compared to formula. The investigators will determine if reflux burden as measured by multichannel intraluminal impedance/esophageal pH monitoring performed for clinical purposes differs between low viscosity conventional formula, medium viscosity commercial blenderized diet, and high viscosity commercial blenderized diet in 45 children receiving conventional formula via gastrostomy. All participants will receive each of the three test diets in random order in a 3-way crossover design. Results of gastric emptying scans will be recorded if done for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-21 years
* G-tube
* Able to tolerate bolus gastric feeds over 30 minutes
* Use of conventional enteral formula
* Undergoing impedance study for clinical purposes

Exclusion Criteria:

* History of allergy or intolerance to any component of the test diets
* History of Nissen fundoplication (participants with suspected or documented unwrapped fundoplication will be eligible for participation)
* Current use of non-invasive pressure support (continuous or bi-level positive airway pressure)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reflux episodes | 4 hours (following feed)
  Number of total reflux episodes (acid and non-acid) by impedance

SECONDARY OUTCOMES:
Full column reflux episodes | 4 hours (following feed)
  Total number of full-column reflux episodes by impedance
Percent of time esophageal pH < 4 | 4 hours after feed
  Percent of time esophageal pH < 4 by impedance
Average height of refluxate | 4 hours after feed
  Average height of refluxate by impedance
Number of symptoms | 4 hours after feed
  Frequency of pulmonary and gastrointestinal symptoms from questionnaires during impedance

OTHER OUTCOMES:
Gastric emptying (percent of ingested contents remaining in stomach at 1 hour) | 1 hour
  Gastric emptying scans by scintigraphy will be analyzed if performed for clinical reasons

CONTACTS AND LOCATIONS:
Overall Officials: Bridget M Hron, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No